CLINICAL TRIAL: NCT05232279
Title: Effect of Testofen on Erectile Function in an Adult Male Population - A Double Blind, Randomised Controlled Trial.
Brief Title: Effect of Testofen on Erectile Function in an Adult Male Population
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESTEF
Record Dates: First submitted 2022-01-18; First posted 2022-02-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Testofen 300mg (Experimental): Testofen in capsule form - taken as a 300mg dosage (2 capsules) once daily for 12 weeks.
  Interventions: Drug: Testofen 300mg
- Testofen 600mg (Experimental): Testofen in capsule form - taken as a 600mg dosage (2 capsules) once daily for 12 weeks.
  Interventions: Drug: Testofen 600mg
- Placebo comparator (Placebo Comparator): The placebo will consist of maltodextrin and will appear identical to the Testofen capsules. The placebo will be administered as per the active treatment - 2 capsules once daily for 12 weeks.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Testofen 300mg — Testofen in capsule form - To be taken as a 300mg dosage (2 capsules) once daily for 12 weeks.
  Arms: Testofen 300mg
Drug: Testofen 600mg — Testofen in capsule form - To be taken as a 600mg dosage (2 capsules) once daily for 12 weeks.
  Arms: Testofen 600mg
Drug: Placebo comparator — The placebo will consist of maltodextrin and will appear identical to the Testofen capsules. The placebo will be administered as per the active treatment - 2 capsules once daily for 12 weeks.
  Arms: Placebo comparator

SUMMARY:
This is a double blind, randomised, placebo-controlled clinical study with a 12-week participation and 3 groups (2 active groups and 1 placebo group) designed to monitor erectile function symptom severity and the effect Testofen may have on improving erectile function, sexual function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged 40-75 years
* Currently in a sexual relationship
* Males with reduced erectile function (Score of <25 on IIEF)
* BMI ≤ 35
* Able to provide informed consent
* Agree not to change current diet and exercise program while enrolled in this trial
* Agree not to undertake another clinical trial while enrolled in this trial

Exclusion Criteria:

* History of prostate surgery and/or trauma
* Receiving/prescribed treatment for erectile dysfunction, including oral medications, vacuum devices, constrictive devices, injections, or urethral suppositories
* Receiving/prescribed treatment to increase/decrease testosterone levels e.g. androgens/anti androgens
* Receiving/prescribed treatment to increase/decrease nitrate or nitric oxide levels
* Unstable or serious illness (e.g. serious mood disorders, neurological disorders such as MS, kidney disease, liver disease, heart conditions, diabetes, hormone production disorders)*
* All current malignancies (excluding BCC) or chemotherapy and/or radiotherapy treatment for malignancy within the previous 2 years
* Receiving/prescribed [e.g., Coumadin or Marevan (warfarin), heparin, dalteparin, enoxaparin) or other anticoagulation therapy (e.g., thromboembolectomy or the use of vena cava filters)
* Active smokers, nicotine use, alcohol, or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in the active or placebo formula
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other related clinical study during the past 1 month

a Any participant reporting having been told by their doctor that they have an under or over production of hormones (e.g., testosterone).

*An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in International Index of Erectile Function (IIEF) questionnaire | Baseline prior to commencement of study product, Week 4, Week 8 and Week 12
  The IIEF is a self-administered questionnaire in which participants will be asked to answer 15 questions relating to erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall sexual satisfaction. Lower scores indicated higher perceived erectile dysfunction
Change in Erection Hardness Score (EHS) | Baseline prior to commencement of study product, Week 4, Week 8 and Week 12
  Participants will be required to assess their erection quality by using the EHS. They will be asked to rate the hardness of their erection on a scale of one to four, with four being the maximal score.

SECONDARY OUTCOMES:
Change in the Ageing Male Symptom (AMS) Questionnaire | Baseline prior to commencement of study product and Week 12
  The Ageing Males' Symptoms scale (AMS) is a self-administered questionnaire that will help assess the symptoms of ageing, often related to androgen decline. As the men in this population are aged between 40 and 75 years, this questionnaire will be used to assess any changes in quality of life.
Change in Derogatis Interview for Sexual Functioning-Self Report (DISF-SR) | Baseline prior to commencement of study product and Week 12
  The DISF-SR is composed of 25 items and examines different aspects of human sexual functioning including sexual cognition and fantasy, sexual arousal, sexual behaviour and experiences, orgasm, and sexual drive and relationship.
Change in cardiovascular health | Baseline prior to commencement of study product and Week 12
  Blood pressure (BP) as measured by automatic blood pressure machine
Change in cardiovascular circulation | Baseline prior to commencement of study product and Week 12
  Doppler flow cytometry of the Femoral artery to assess circulation
Change in height in anthropometry measurements | Baseline prior to commencement of study product and Week 12
  Height as measured by stadiometer in centimeters
Change in weight in anthropometry measurements | Baseline prior to commencement of study product and Week 12
  Weight as measured by digital scales in kilograms
Change in waist circumference in anthropometry measurements | Baseline prior to commencement of study product and Week 12
  Waist circumference as measured by tape in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD information will be shared